CLINICAL TRIAL: NCT03342547
Title: Genome-wide CRISPR Screen for Host Factors Associated With Norovirus Infections in Stem Cell-derived Human Intestinal Enteroid Model
Brief Title: Identification of Host Factors of Norovirus Infections in Mini-Gut Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHAN CHI WAI, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MIC_CHAN_GRF_17_18_v1_20160930
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Gastrointestinal Infection
Keywords: Norovirus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intestinal stem cell-derived enteroids (Experimental): Duodenal biopsy samples and saliva will be collected from participants and then processed in laboratory to generate intestinal stem cell-derived enteroids.
  Interventions: Procedure: Duodenal biopsy; Procedure: Saliva

INTERVENTIONS:
Procedure: Duodenal biopsy — Two duodenal biopsy samples will be collected from each participant
Procedure: Saliva — Saliva (1-2 mL) will be collected from each participant for secretor status testing

SUMMARY:
The primary objective in this study is to establish a list of host cellular proteins that mediate norovirus infection.

Norovirus is one of the most common pathogens attributed to diarrheal diseases from unsafe food. It is also the primary cause of mortality among young children and adults in foodborne infections. Norovirus is not just a foodborne burden. In a recent meta-analysis, norovirus accounts for nearly one-fifth of all causes of (including person-to-person transmission) acute gastroenteritis in both sporadic and outbreak settings and affects all age groups. Undoubtedly, norovirus is of paramount public health concern in both developed and developing countries. Research efforts to better understand norovirus pathobiology will be necessary for targeted intervention.

From Middle East respiratory syndrome coronavirus to Zika virus, efforts to identify host factors important for mediating virus infection has always been a research priority. Such information will shed light on potential therapeutic targets in antiviral intervention. Norovirus virus-host interaction studies have been hampered by the lack of a robust cell culture model in the past 20 years. In 2016, norovirus has finally been successfully cultivated in a stem cell-derived three-dimensional human gut-like structure called enteroid or mini-gut.

In this study, intestinal stem cells will be isolated from duodenal biopsies collected from participants, followed by differentiation into mini-guts. Genome-wide genetic screening for host essential and restrictive factors will be performed on infected mini-guts by knockout CRISPR and gain-of-function CRISPR SAM, respectively. Shortlisted candidates will undergo preliminary functional validation in cell lines. These data will provide insights into potential therapeutic targets against norovirus infection.

DETAILED DESCRIPTION:
Study design and overview - This is a laboratory-based study. The investigators plan to establish a list of host cellular proteins regulating norovirus infection. Methods will include establishment of patient-specific stem cell-derived human intestinal enteroids as an infection model and genome-wide CRISPR and CRISPR SAM genetic screens upon infections of two norovirus genotypes.

***Establishment of human intestinal enteroid model***

1. Duodenal biopsies and saliva collection - After obtaining IRB-approved informed consent, two duodenal biopsy samples will be obtained from each participant undergoing upper gastrointestinal endoscopy without contraindications for biopsy sampling, such as participants on anti-coagulation or with other causes of bleeding diathesis. Biopsy samples will be immersed in ice-cold 1xPBS and transported immediately to the laboratory within 30 minutes for further processing. In addition, saliva (1-2 mL) will be collected from each participant for secretor status testing by ELISA.
2. Isolation of crypt stem cells and differentiation - Upon arrival, biopsy samples will first be chopped into smaller pieces. Intestinal crypt cells will be isolated by repeated washing and incubation with 1x Complete Chelating solution (1xCCS) and EDTA buffer. Supernatant containing crypt cells will then be grown in Matrigel containing complete medium with growth factors (CMGF+) (Wnt 3 and Rspo-1 conditioned media, Noggin, A83, B27, EGF, N2, n-acetylcysteine, gastrin, nicotinamide, and SB202190). Budding crypts will then be incubated in differentiation medium (CMGF+, excluding Wnt 3 conditioned medium, SB202190 and nicotinamide as well as having reduced amount of Rspo-1 conditioned medium and Noggin). Formation of three-dimensional gut-like enteroids will be monitored daily.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or above
* Prospective outpatients undergoing gastrointestinal endoscopy for symptoms of dyspepsia in the Endoscopy Unit of the Prince of Wales Hospital, Shatin, Hong Kong, China
* Able and willing to provide informed written consent

Exclusion Criteria:

* Use of anti-coagulants and/or aspirin that may have increased risk of bleeding
* History of bleeding diathesis
* Contraindications for biopsy sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-04-18 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Establishment of human intestinal stem cell-derived enteroids | An average of three months
  Viability of enteroids as determined by microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Wai Chan, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Endoscopy Centre, Prince of Wales Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided